CLINICAL TRIAL: NCT05263193
Title: Retrospective Data Collection of Pediatric Patients With Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP) Treated With Caplacizumab
Brief Title: Retrospective Study on Caplacizumab-treated Pediatric Patients With Immune-mediated Thrombocytopenic Purpura (iTTP)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17325
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Immune-mediated Thrombocytopenic Purpura
MeSH Terms: interventions — caplacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Caplacizumab — as in real world practice
  Other Names: Cablivi®

SUMMARY:
The purpose of this multi-country, retrospective data collection study (chart review) is to describe the effectiveness and safety of caplacizumab in pediatric patients with iTTP.

DETAILED DESCRIPTION:
Pediatric patients who received caplacizumab will be identified for enrollment in the chart review. The eligibility period starts on August 30, 2018 in the United Kingdom (UK) and France and February 6, 2019 for the United States (US).

Data collection is fully retrospective and will be anchored to the patient's index event date. The index event date is defined as the date the patient initiated caplacizumab treatment. The study period begins at the index date and ends at the earliest date of chart abstraction initiation, 12 weeks after last dose of caplacizumab treatment, date of death, or loss to follow-upwhich ever comes first .

ELIGIBILITY:
Inclusion Criteria:

* Patient's aged ≤18 years at start of caplacizumab treatment initiation
* Patient has a diagnosis of iTTP documented in the medical records
* Patient was treated with caplacizumab within the eligibility period

Exclusion Criteria:

* Patient declined use of data for study (where local regulations require patient notification of planned study)
* Patient's medical chart is missing or not retrievable

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with Immune-mediated Thrombotic Thrombocytopenic Purpura treated with Caplacizumab
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Platelet count response | From index date up to 12 weeks after last dose of caplacizumab
  defined as time from caplacizumab initiation to initial platelet count ≥ 150×109/L with subsequent stop of daily plasma exchange (PE) within 5 days
Proportion of subjects with refractory iTTP | From index date up to 12 weeks after last dose of caplacizumab
  defined as lack of doubling of platelet count after four days of caplacizumab treatment and a lactate dehydrogenase (LDH) level that remained above the upper limit of normal (ULN) range
Proportion of subjects with recurrent disease | From index date up to 12 weeks after last dose of caplacizumab
  Proportion of subjects with iTTP exacerbation (defined as recurrence within 30 days after last PE) and Proportion of subjects with iTTP relapse (defined as recurrence more than 30 days after last PE)
Time to normalization of organ damage marker levels | From index date up to 12 weeks after last dose of caplacizumab
  Defined asLDH ≤ 2 x ULN, Serum creatinine ≤ 1 x ULN, Cardiac troponin I ≤ 1 x ULN
Total duration of hospitalization stays | From index date up to 12 weeks after last dose of caplacizumab
Duration of intensive care unit (ICU) stay | From index date up to 12 weeks after last dose of caplacizumab
Duration of therapeutic PE | From index date up to 12 weeks after last dose of caplacizumab
Proportion of patients achieving clinical response | From index date up to 12 weeks after last dose of caplacizumab
  defined as a normal platelet countand LDH < 2 ULN for at least 48 hours following initial normalization or response of platelet count
Time to ADAMTS13 activity ≥ 20% | From index date up to 12 weeks after last dose of caplacizumab
  where available and feasible
Number of participants with Adverse event | From index date up to 12 weeks after last dose of caplacizumab
  including serious adverse events

SECONDARY OUTCOMES:
Treatment pattern of caplacizumab therapy | From index date up to 12 weeks after last dose of caplacizumab
  Dosing and duration
Types and duration of concomitant medications | From index date up to 12 weeks after last dose of caplacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org